CLINICAL TRIAL: NCT01891318
Title: Neoadjuvant Radiosurgery for Resectable Brain Metastases: Phase I/II Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7312
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Tumors Metastatic to Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (radiosurgery, surgery) (Experimental): Patients undergo radiosurgery on day 0. Within 2 weeks, patients undergo surgical resection.
  Interventions: Radiation: radiosurgery; Procedure: therapeutic conventional surgery; Procedure: quality-of-life assessment

INTERVENTIONS:
Radiation: radiosurgery — Undergo radiosurgery
  Other Names: radiation surgery
Procedure: therapeutic conventional surgery — Undergo surgical resection
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This Phase I/II trial studies the ability to stop brain metastases from coming back after treatment with radiosurgery followed by surgical resection. It will also evaluate the side effects of these combined treatments and help determine the best radiosurgery dose. Radiosurgery focuses the x-rays directly to the tumor and cause less damage to the normal tissue in the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety (risk of acute and long-term toxicities) of neoadjuvant radiosurgery at escalating doses followed by surgical resection of brain metastases. (Phase I)

II. To determine the local control of brain metastases treated with neoadjuvant radiosurgery followed by surgical resection. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the rate of distant brain failure when brain metastases are managed with neoadjuvant radiosurgery followed by surgical resection.

II. To estimate the rate of salvage surgery, whole brain radiation therapy (WBRT), or stereotactic radiosurgery (SRS) for participants treated with neoadjuvant radiosurgery followed by surgical resection.

III. To determine the rate of radiation necrosis/steroid dependency. IV. To determine the radiobiologic impact of neoadjuvant radiosurgery for resected brain metastases.

OUTLINE: This is a phase I, dose-escalation study of radiosurgery followed by a phase II study.

The following outcomes were removed from the protocol in an amendment:

* Changes in neurocognitive function as measured by the Hopkins Verbal Learning Test (HVLT), Controlled Oral Word Association (COWA) & Trailmaking Test B, and Trailmaking Test A
* QOL measured by FACT-BR and EORTC-QLQ30

ELIGIBILITY:
Inclusion Criteria:

* Have a prior histologic diagnosis of cancer other than small cell lung cancer, lymphoma, and germ cell histologies
* Magnetic resonance imaging (MRI) evidence of 1-4 brain metastases, with at least one lesion > 20 mm and ≤ 50 mm in maximal diameter and determined to be appropriate for SRS and gross total resection; all other brain metastases are appropriate for SRS
* Patient can have prior SRS to lesions other than the one planned for neoadjuvant SRS and resection
* Patient must have a Karnofsky performance score of ≥ 70

Exclusion Criteria:

* Patient deemed medically unfit to undergo surgical resection of brain metastasis
* Prior whole brain radiotherapy
* Patient with contraindication for imaging with MRI
* Inability to participate in study activities due to physical or mental limitations
* Inability or unwillingness to return for all the required follow-up visits
* At the time of planning, unable to deliver 10 Gray (Gy) or less to optic nerve/chiasm
* Tumor located in the brainstem
* Imaging or cytologic evidence of leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-07-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Day 0
  MTD of radiosurgery determined by dose-limiting toxicities graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 (Phase I)
Proportion of participants without local failure (Phase II) | Up to 3 years
  Local control of brain metastases, as measured by proportion of participants without local failure (Local failure is tumor progression of the metastasis treated on the study)
  (Phase II)
  The Kaplan-Meier method will be used.

SECONDARY OUTCOMES:
Proportion of participants with distant brain failure | Up to 3 years
  Rate of distant brain failure, defined as progression of brain metastases outside of the brain metastasis treated on study. The Kaplan-Meier method will be used.
Rate of radiation necrosis/steroid dependency | Up to 3 years
  Rate of radiation necrosis/steroid dependency
Rate of salvage treatment | Up to 3 years
  Number of patients that have any salvage treatment, including surgery, stereotactic radiosurgery (SRS), or whole brain radiation therapy (WBRT)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Murphy, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio